CLINICAL TRIAL: NCT00206245
Title: A Randomised, Double-blind, Multicentre Dose-finding Phase IIb Study for up to 8 Weeks' Treatment With AZD0865 25, 50, 75 mg and Esomeprazole 40 mg, Given Orally Once Daily for the Healing of Erosive Esophagitis in Adult Subjects With GERD With Erosive Esophagitis According to the LA Classification in Adult Subjects.
Brief Title: A Dose-finding Phase IIb Study With AZD0865 and Esomeprazole in GERD Patients With Erosive Esophagitis.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D9770C00012
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2013-01

CONDITIONS: GERD With Erosive Esophagitis
Keywords: GERD with erosive esophagitis
MeSH Terms: interventions — AZD0865

INTERVENTIONS:
Drug: AZD0865

SUMMARY:
The primary objective is to compare the efficacy between three doses of AZD0865 (25, 50 and 75 mg).

The secondary objectives are to compare the efficacy between the three doses of AZD0865 and esomeprazole 40 mg and to evaluate the safety and tolerability of AZD0865.

ELIGIBILITY:
Inclusion Criteria:

* Identification of their main symptom as heartburn defined as a burning feeling behind the breastbone.
* Have at least a 6-month history of heartburn and at least 4 days of episodes of heartburn with at least overall moderate intensity during the last 7 days prior to visit 1.
* Erosive esophagitis according to LA classification Grade A, B, C or D, at the visit 1 endoscopy.
* Have provided Informed consent.

Exclusion Criteria:

Subjects with current or historical evidence of the following conditions are excluded from the study:

* Esophageal stricture.
* Primary esophageal motility disorder(s), i.e. diffuse esophageal spasm, achalasia.
* Systemic Sclerosis (scleroderma).
* Irritable Bowel Syndrome (IBS), i.e. upper abdominal discomfort or pain that in the opinion of the Investigator is likely to be due to IBS or fulfilling two or more of the criteria: relieved by defecation, associated with change in frequency of stools, associated with change in form (appearance) of stools.
* Inflammatory bowel disease.
* Zollinger-Ellison syndrome.
* Gastric ulcer, duodenal ulcer or duodenal erosions within the last 3 months

Subjects with i) history of significant or ii) current significant or unstable:

* Cardiovascular diseases or cardiac chest pain.
* Cerebrovascular diseases, such as cerebral ischemia, infarction, haemorrhage, or embolus.
* Diabetes mellitus. Stable diabetes controlled on diet, oral agents or insulin is acceptable.
* Pulmonary, renal, pancreatic or liver diseases or any other serious disease as judged by the investigator to interfere with the evaluation of the current study.
* Malignant disease (except for minor superficial skin disease).
* Generalised bleeding disorders.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1400
Dates: Start 2004-05; Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Healing of erosive esophagitis at 4 weeks.

SECONDARY OUTCOMES:
Healing of erosive esophagitis at 2 and 8 weeks.
The Quality of Life in Reflux and Dyspepsia (QOLRAD).
Patient-reported symptoms.
Investigator-reported symptoms.
Population pharmacokinetics (PK). Area under the concentration-time curve (AUC) and the oral clearance calculated by dose/AUC (CL/F).
pH monitoring.
Histology.
Safety (Adverse events, Laboratory variables, BP, pulse, ECG and physical examination).

CONTACTS AND LOCATIONS:
Locations (202):
- United States (77):
  - Research Site, Alabaster, Alabama
  - Research Site, Huntsville, Alabama
  - Research Site, Tucson, Arizona
  - Research Site, North Little Rock, Arkansas
  - Research Site, Anaheim, California
  - Research Site, Cypress, California
  - Research Site, Garden Grove, California
  - Research Site, Lancaster, California
  - Research Site, Los Angeles, California
  - Research Site, Mission Hills, California
  - Research Site, Orange, California
  - Research Site, Rancho Cucamonga, California
  - Research Site, San Diego, California
  - Research Site, Torrance, California
  - Research Site, Wheat Ridge, Colorado
  - Research Site, Manchester, Connecticut
  - Research Site, Davie, Florida
  - Research Site, Gainesville, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Jupiter, Florida
  - Research Site, Miami, Florida
  - Research Site, Ocoee, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Zephyrhills, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Austell, Georgia
  - Research Site, Conyers, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Moline, Illinois
  - Research Site, Rockford, Illinois
  - Research Site, Clive, Iowa
  - Research Site, Overland Park, Kansas
  - Research Site, Metairie, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, Annapolis, Maryland
  - Research Site, Baltimore, Maryland
  - Research Site, Hollywood, Maryland
  - Research Site, Laurel, Maryland
  - Research Site, Towson, Maryland
  - Research Site, Picayune, Mississippi
  - Research Site, Jefferson City, Missouri
  - Research Site, Kansas City, Missouri
  - Research Site, Butte, Montana
  - Research Site, Willingboro, New Jersey
  - Research Site, Charlotte, North Carolina
  - Research Site, Elkin, North Carolina
  - Research Site, Fayetteville, North Carolina
  - Research Site, Greensboro, North Carolina
  - Research Site, Greenville, North Carolina
  - Research Site, High Point, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Canton, Ohio
  - Research Site, Guthrie, Oklahoma
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Duncansville, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Anderson, South Carolina
  - Research Site, Georgetown, South Carolina
  - Research Site, Mt. Pleasant, South Carolina
  - Research Site, Simpsonville, South Carolina
  - Research Site, Bristol, Tennessee
  - Research Site, Chattanooga, Tennessee
  - Research Site, Jackson, Tennessee
  - Research Site, Knoxville, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Ogden, Utah
  - Research Site, Salt Lake City, Utah
  - Research Site, Christiansburg, Virginia
  - Research Site, Norfolk, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Spokane, Washington
  - Research Site, Tacoma, Washington
  - Research Site, Milwaukee, Wisconsin
- Canada (16):
  - Research Site, Abbotsford, British Columbia
  - Research Site, Vancouver, British Columbia
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Halifax, Nova Scotia
  - Research Site, Guelph, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, Mississauga, Ontario
  - Research Site, North York, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Thornhill, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Lévis, Quebec
  - Research Site, Longueuil, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Saskatoon, Saskatchewan
- Denmark (14):
  - Research Site, Aalborg
  - Research Site, Århus C
  - Research Site, Birkerød
  - Research Site, Esbjerg
  - Research Site, Herning
  - Research Site, Holbæk
  - Research Site, Hvidovre
  - Research Site, Kolding
  - Research Site, København K
  - Research Site, København NV
  - Research Site, Odense
  - Research Site, Randers
  - Research Site, Vejle
  - Research Site, Viborg
- Finland (8):
  - Research Site, Espoo
  - Research Site, Helsinki
  - Research Site, Lahti
  - Research Site, Mikkeli
  - Research Site, Pori
  - Research Site, Tampere
  - Research Site, Turku
  - Research Site, Vantaa
- France (16):
  - Research Site, Alès
  - Research Site, Angers
  - Research Site, Beausoleil
  - Research Site, Bordeaux
  - Research Site, Caen
  - Research Site, Cannes La Bocca
  - Research Site, Choisy-le-Roi
  - Research Site, Dreux
  - Research Site, Hazebrouck
  - Research Site, Issoire
  - Research Site, Marseille
  - Research Site, Narbonne
  - Research Site, Paris
  - Research Site, Saint-Quentin
  - Research Site, Talence
  - Research Site, Vitry-sur-Seine
- Germany (14):
  - Research Site, Berlin
  - Research Site, Celle
  - Research Site, Cologne
  - Research Site, Dresden
  - Research Site, Görlitz
  - Research Site, Leipzig
  - Research Site, Ludwigshafen
  - Research Site, Magdeburg
  - Research Site, Mainz
  - Research Site, München
  - Research Site, Oelde
  - Research Site, Potsdam
  - Research Site, Ribnitz-Damgarten
  - Research Site, Wolmirstedt
- Italy (10):
  - Research Site, Bologna
  - Research Site, Brescia
  - Research Site, Genova
  - Research Site, Mestre
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Palermo
  - Research Site, Parma
  - Research Site, Pisa
  - Research Site, Roma
- Norway (10):
  - Research Site, Bergen
  - Research Site, Bodø
  - Research Siteq, Drammen
  - Research Site, Gjøvik
  - Research Site, Levanger
  - Research Site, Nesttun
  - Research Site, Oslo
  - Research Site, Stavanger
  - Research Site, Tromsø
  - Research Site, Trondheim
- Sweden (14):
  - Research Site, Karlskrona
  - Research Site, Kristianstad
  - Research Site, Kungälv
  - Research Site, Malmo
  - Research Site, Mora
  - Research Site, Nyköping
  - Research Siteq, Östersund
  - Research Site, Säffle
  - Research Site, Skövde
  - Research Site, Stockholm
  - Research Site, Sundsvall
  - Research Site, Täby
  - Research Site, Varberg
  - Research Site, Värnamo
- United Kingdom (23):
  - Research Site, Ashford
  - Research Site, Atherstone
  - Research Site, Cambridge
  - Research Site, Cheltenham
  - Research Site, Coventry
  - Research Site, Derby
  - Research Site, Dundee
  - Research Site, Dunfermline
  - Research Site, Epsom
  - Research Site, Glasgow
  - Research Site, Hamilton
  - Research Site, Kent
  - Research Site, Lancaster
  - Research Site, Manchester
  - Research Site, Slough
  - Research Site, Somerset
  - Research Site, Stafford
  - Research Site, Stockport
  - Research Site, Telford
  - Research Site, Torquay
  - Research Site, West Bromwich
  - Research Site, West Yorks
  - Research Site, Woking

REFERENCES:
- [Derived] Kahrilas PJ, Persson T, Denison H, Wernersson B, Hughes N, Howden CW. Predictors of either rapid healing or refractory reflux oesophagitis during treatment with potent acid suppression. Aliment Pharmacol Ther. 2014 Sep;40(6):648-56. doi: 10.1111/apt.12877. Epub 2014 Jul 15. PMID 25039978
- [Derived] Kahrilas PJ, Jonsson A, Denison H, Wernersson B, Hughes N, Howden CW. Impact of regurgitation on health-related quality of life in gastro-oesophageal reflux disease before and after short-term potent acid suppression therapy. Gut. 2014 May;63(5):720-6. doi: 10.1136/gutjnl-2013-304883. Epub 2013 Jul 5. PMID 23831734